CLINICAL TRIAL: NCT02120170
Title: The Effect of Prophylactic Clip Application for Colon Polypectomy in Patients With Anticoagulation: Prospective Randomized Controlled Trial
Brief Title: Prophylactic Clip Application for Colon Polypectomy in Patients With Anticoagulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Gun, Kim. M.D., Ph.D., Associate professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIPO
Record Dates: First submitted 2014-03-27; First posted 2014-04-22 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Colon Polyp
Keywords: Hemoclip, Heparin bridging therapy, colon polypectomy, warfarin
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemoclipping during colon polypectomy for all lesion (Active Comparator): The enrolled patients of group 1 will be performed hemoclipping for all polypectomy lesion irrespective of the presence of immediate bleeding.
  Interventions: Procedure: Colon polypectomy
- No hemoclipping if there were no bleeding during polypectomy (No Intervention): The patients of group 2 will be performed hemoclipping only for the immediate bleeding during colon polypectomy

INTERVENTIONS:
Procedure: Colon polypectomy
  Arms: Hemoclipping during colon polypectomy for all lesion

SUMMARY:
There have been very limited evidence about the bleeding complication during colon polypectomy for the patients taking warfarin.

This study is aimed to analyse the effect of prophylactic hemo-clipping during colon polypectomy for the patients with warfarin consumption.

The enrolled subjects are the patients who take warfarin for high thromboembolism risk and should take heparin bridging therapy during colon polypectomy instead of temporary stopping warfarin. The investigators will randomize into two groups; the patient enrolled into group 1 will be performed hemoclipping for all polypectomy lesion irrespective of the presence of immediate bleeding. And the patients enrolled into group 2 will be performed hemoclipping only for the lesion of immediate bleeding during colon polypectomy.

The primary endpoint is to compare the rate of delayed bleeding between two groups.

DETAILED DESCRIPTION:
The American guideline have recommended that if the patient with low risk of thromboembolism, warfarin consumption can be quit 3~5 days before colon polypectomy and resume within 24 hours after polypectomy. However, if the patient were high risk of thromboembolism, the patient should take heparin bridging therapy during temporal quit of warfarin consumption for colon polypectomy. There have been very limited evidences about the bleeding complication during colon polypectomy for the patients with warfarin taking.

Moreover, there have been lack of evidence that how to prevent the bleeding complication in the patients with high risk of thromboembolism who should take heparin bridging therapy during temporal stopping of warfarin for colon polypectomy.

This study is aimed to analyse the effect of prophylactic hemo-clipping during colon polypectomy for the patients with warfarin consumption.

The investigators will enroll the subjects who should take heparin bridging therapy (quit warfarin 3~5 days before colon polypectomy and check the INR, if the INR <2, heparin or low molecular heparin should be start. If the INR <1.5 on the day before colon polypectomy, the patient will undergo bowel preparation and colon polypectomy. Warfarin will resume within 24 hour after polypectomy) after quit warfarin for during colon polypectomy over 19 years old.

Exclusions are as follow; patients who don't have to take bridging heparin therapy after quit warfarin, patients have low a platelet count (<80,000/mm3), patients who take anti-platelet agents, patients who have GI malignancies. The investigators will randomize into two groups; the patient enrolled into group 1 will be performed hemoclipping for all polypectomy lesion irrespective of the presence of immediate bleeding. And the patients enrolled into group 2 will be performed hemoclipping only for the lesion of immediate bleeding during colon polypectomy. Including polyps for colon polypectomy are 6~ 20 mm size and polypectomy procedure is defined as EMR after injection with blended electrical current.

The lesion which immediate bleeding is occurred during the polypectomy will be performed hemoclipping irrespective of group and will not be counted as delayed bleeding even though delayed bleeding is occurred on this lesion.

The primary endpoint is to compare the rate of delayed bleeding between two groups. The secondary endpoint is to analyse the effect of hemoclipping for immediate bleeding.

This study will be performed during 3 years after 1st patient enrollment and the target size of enrollment is 356 (176 in each group).

ELIGIBILITY:
Inclusion Criteria:

* subjects who should take heparin bridging therapy after quit warfarin 3~5 days before colon polypectomy because of high risk of thromboembolism - AF with valvular disease, AF with mechanical valve, AF with CHF, EF <35%, AF with previous thromboembolism, AF with DM and HTN, AF with old age(>75),

Exclusion Criteria:

* patients who don't have to take bridging heparin therapy after quit warfarin, patients have low a platelet count (<80,000/mm3), patients who take anti-platelet agents, patients who have GI malignancies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with delayed bleeding | Bleeding within 30 days after colon polypectomy
  The primary endpoint is to compare the rate of delayed bleeding between two groups.

SECONDARY OUTCOMES:
Number of successful bleeding control after hemoclipping for immediate bleeding in the patients with warfarin. | Bleeding during the procedure
  The secondary endpoint is to analyse the effect of hemoclipping for immediate bleeding and will be measured as successful hemostasis rate of hemoclipping. There has limited evidence about the efficacy of hemoclipping for the immediate bleeding during colon polypectomy in the patients with anticoagulation

OTHER OUTCOMES:
Cut-off value of resuming timing of warfarin after colon polypectomy | Within 1 week after polypectomy
  The guideline recommended warfarin resuming within 24 hours after colon polypectomy, But there is very limited evidence about safe timing of warfarin resuming regarding the bleeding complication.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Gun Kim, MD.,PhD., Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Hospital, Seoul, Seoul, South Korea